CLINICAL TRIAL: NCT05658562
Title: A Phase I/II Open-Label Study of MT-2111 in Patients With Relapsed/Refractory DLBCL
Brief Title: A Study of MT-2111 in Patients With Relapsed/Refractory DLBCL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-2111-A-101
Record Dates: First submitted 2022-11-07; First posted 2022-12-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MT-2111 dosing regimen (Experimental)
  Interventions: Drug: MT-2111

INTERVENTIONS:
Drug: MT-2111 — i.v. infusion
  Other Names: Loncastuximab tesirine

SUMMARY:
[Phase I part] To investigate the safety, tolerability, and pharmacokinetics of MT-2111 monotherapy in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). In addition, the dose to be used in the Phase II part will be confirmed.

[Phase II part] To evaluate the efficacy of MT-2111 monotherapy in patients with relapsed/refractory DLBCL. In addition, the safety and pharmacokinetics will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed pathologically with DLBCL, NOS, DLBCL transformed from indolent B-cell lymphoma, or high-grade B-cell lymphoma with DLBCL morphology and with MYC and BCL2 and/or BCL6 rearrangements, based on the 2017 WHO classification.
* Patients with relapsed or refractory disease despite 2 or more prior systemic therapies.
* Japanese patients aged ≥ 18 years at the time of informed consent. For Japanese subjects, it should be confirmed that the parents who are related by blood to the subject must be Japanese.
* Patients who have a lesion that can be assessed for staging and evaluated for response according to the Lugano criteria (2014). A lesion that has received radiotherapy as the most recent treatment will be considered as a measurable lesion only when progression has been documented following completion of the radiotherapy.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at screening.

Exclusion Criteria:

* Patients with a pathological diagnosis of Burkitt's lymphoma.
* Patients with bulky disease with the longest dimension of ≥ 10 cm.
* Patients with a history or complication of post-transplant lymphoproliferative disorders.
* Patients with lymphoma with active central nervous system involvement at the time of screening, including leptomeningeal disease.
* Patients complicated with other active malignancies or patients with a history of other malignancies within 3 years before informed consent. However, the following are exceptional:

  * Non-melanoma skin cancer
  * Non-metastatic prostate cancer
  * Cervical carcinoma in situ
  * Ductal carcinoma in situ or lobular carcinoma in situ
* Patients with clinically significant third space fluid accumulation (e.g., ascites requiring drainage or pleural effusion requiring drainage or associated with shortness of breath).
* Patients who underwent autologous hematopoietic stem cell transplantation (AHSCT) within 30 days prior to the start of study drug administration (Cycle 1 Day 1).
* For the Phase I part, patients with prior allogeneic stem cell transplantation (Allo-HSCT) before the start of study drug administration (Cycle 1 Day 1). For the Phase II part, patients undergoing Allo-HSCT within 60 days prior to the start of study drug administration (Cycle 1 Day 1).
* Patients who had a positive HIV antigen-antibody test or HIV antibody test.
* Patients positive for HBs antigen, HBc antibody, or HBs antibody. However, patients who meet any of the following are eligible:

  * The patient's HBs antibody positivity is clearly due to vaccination.
  * Patients who are positive for HBs antibody and/or HBc antibody with HBV-DNA not detected and agree to undergo HBV-DNA tests once a month from the start of study drug administration to at least 12 months after the completion of study drug administration.
* Patients positive for HCV antibody. However, patients with negative HCV-RNA are eligible.
* Patients who received anticancer therapy during the following periods prior to the start of study drug administration (Cycle 1 Day 1).

  * Cytotoxic chemotherapy: within 14 days.
  * Antibody therapy: within 5 half-lives or 14 days, whichever is longer (including monoclonal antibody preparations, radioimmunoconjugates, or antibody-drug conjugates). Within 14 days for rituximab, anti-CD3/CD20 bispecific antibody.
  * Radiotherapy: within 14 days
  * CAR-T therapy: within 100 days
  * Other anticancer therapy: within 14 days
* Patients who received treatment with any other investigational product within 14 days prior to the start of study drug administration (Cycle 1 Day 1). However, for the Phase I part, patients who received any other investigational product within 14 days or 5 half-lives, whichever is longer, before the start of study drug administration (Cycle 1 Day 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) by independent central review | From the date of first dose of study treatment until all participants completed treatment period or discontinued treatment (Up to 12 months)

SECONDARY OUTCOMES:
Duration of response (DOR) | The time from the date of first observation of complete response (CR) or partial response (PR) until progressive disease (PD) or death in patients with CR or PR observed (Up to 48 months)
Complete response rate (CRR) | From the date of first dose of study treatment until all participants completed treatment period or discontinued treatment (Up to 12 months)
Overall survival (OS) | The time from the date of first dose until death regardless of the occurrence of intercurrent event (Up to 48 months)
Progression-free survival (PFS) | The time from the date of first dose until PD or death (Up to 48 months)
Relapse-free survival (RFS) | The time from the date of first observation of CR until PD or death in patients with CR observed (Up to 48 months)
Adverse events and adverse drug reactions | From the start of premedication until 15 weeks after the last dose of the study drug or until the start of new anticancer therapy, whichever comes first.
Eastern Cooperative Oncology Group (ECOG) Performance Status | Screening to end of treatment (up to 30 days after the last dose) or data cut off
  ECOG (Eastern Cooperative Oncology Group) Performance Status is scored on a 6-point scale where higher scores indicate a worse outcome.
Body weight | Screening to end of treatment (up to 30 days after the last dose) or data cut off
12-lead electrocardiogram (heart rate) | Screening to end of treatment (up to 30 days after the last dose) or data cut off
12-lead electrocardiogram [RR, PR, QRS, QT (QTcF)] | Screening to end of treatment (up to 30 days after the last dose) or data cut off
12-lead electrocardiogram (presence or absence of abnormal findings) | Screening to end of treatment (up to 30 days after the last dose) or data cut off
Serum drug concentration | Please refer to the description above
  [Phase 1 part] Cycle 1 [each cycle is 3 weeks (21 days) in duration]: Day 1, 2, 5, 8 and 15, Cycle 2: Day 1, 2, 8 and 15, Cycle 3: Day 1 and 8, odd number Cycle: Day 1,end of treatment (EOT)*, and 15 weeks after EOT* [Phase 2 part] Cycle 1 and 2: Day 1, 8 and 15, odd number Cycle : Day 1, EOT*, and15 weeks after EOT*
  *: After the decision to discontinue treatment with study drug and prior to the start of any new anticancer therapy, the scheduled evaluations will be performed preferably 30 days after the last dose of study drug.
  One cycle is 3 weeks (21 days) in duration.
  *: After the decision to discontinue treatment with study drug and prior to the start of any new anticancer therapy, the scheduled evaluations will be performed preferably 30 days after the last dose of study drug.
Anti-drug antibodies (including neutralizing antibodies) | Please refer to the description above.
  [Phase 1 part] Cycle 1 [each cycle is 3 weeks (21 days) in duration]: Day 1 and 15, Cycle 2: Day 1, odd number Cycle: Day 1, end of treatment (EOT)*, and 15 weeks after EOT* [Phase 2 part] Cycle 1: Day 1 and 15, Cycle 2: Day 1, odd number Cycle : Day 1, EOT*, and 15 weeks after EOT*
  *: After the decision to discontinue treatment with study drug and prior to the start of any new anticancer therapy, the scheduled evaluations will be performed preferably 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (23):
- Japan (23):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kyushu Cancer Center, Fukuoka, Fukuoka
  - Aso Iizuka Hospital, Iizuka-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gunma Prefectural Cancer Center, Ota-shi, Gunma
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki, Nagasaki
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Medical Research Institute KITANO HOSPITAL, PIIF Tazuke-kofukai, Osaka, Osaka
  - Shimane University Hospital, Izumo-shi, Shimane
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Disaster Medical Center, Tachikawa-shi, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
When requested by a qualified researcher in the field of science or medicine, Tanabe Pharma Corporation will share clinical trial data that was collected from individual patients in a clinical trial with that researcher after a review committee of experts determines that such sharing is appropriate.
  Access Criteria: Please refer to the following link for conditions and limitations for sharing data.
  URL: https://www.tanabe-pharma.com/en/develop/protocol.html